CLINICAL TRIAL: NCT03975075
Title: Biofeedback Treatment of Anxiety Associated With Chronic Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Hospital (Other)
Responsible Party: Principal Investigator, Kimberley R Monden, Senior Principal Investigator, University of Minnesota
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 594559
Record Dates: First submitted 2019-05-16; First posted 2019-06-05 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Spinal Cord Injuries; Anxiety; Stress; Tetraplegia
MeSH Terms: conditions — Spinal Cord Injuries; Anxiety Disorders; Quadriplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback (Experimental): Participants (n=15) will undergo 30 minutes of self-administered 1-channel (ECG) physiological monitoring at home using the Mindfield eSense Pulse twice a week for four weeks (eight sessions in total). The biofeedback training session will be conducted using the eSense Pulse smartphone application. Participants will receive further instruction explaining how physiological information will be displayed and used as a means of training to induce a relaxed state while receiving real time feedback. Participants will be instructed on using controlled breathing to assist with reaching this relaxed state. Prior to each training session, the Study Coordinator will meet with the participant via Zoom to virtually assist with setup. Following each training session, participants will respond to questionnaires over the phone.
  Interventions: Behavioral: Psychophysiological monitoring; Behavioral: Biofeedback training
- Control Group (Active Comparator): Participants (n=15) will undergo 30 minutes of self-administered 1-channel (ECG) physiological monitoring at home using the Mindfield eSense Pulse twice a week for four weeks (eight sessions in total). Participants will be provided with the following instructions: "You will be monitored with this equipment for 30 minutes. During this time frame, please try to limit movement and conversation as much as possible." Prior to each training session, the Study Coordinator will meet with the participant via Zoom to virtually assist with setup. Following each training session, participants will respond to questionnaires over the phone.
  Interventions: Behavioral: Psychophysiological monitoring

INTERVENTIONS:
Behavioral: Psychophysiological monitoring — 30 minutes of one channel (ECG) physiological monitoring with Mindfield eSense Pulse.
Behavioral: Biofeedback training — Traditional resonance frequency training with the Mindfield eSense Pulse smartphone application. Using visual feedback of real time parameters of HRV and the use of controlled breathing, participants are trained to reach a relaxed state.
  Arms: Biofeedback

SUMMARY:
The purpose of this research is to test the feasibility of an intervention using biofeedback to treat stress and anxiety among individuals with tetraplegia.

The expected duration of participation in this study is about 5 hours over the course of about 5 weeks. Participants will be randomly assigned to either a biofeedback training intervention or a control group. After completing questionnaires, participants will undergo physiological monitoring for the purpose of measuring heart rate and breathing. Those assigned to the biofeedback group will undergo 20 minutes of physiological monitoring while also participating in biofeedback training twice a week for 4 weeks (8 sessions) from home. Those assigned to the control group will undergo 20 minutes of physiological monitoring twice a week for 4 weeks (8 sessions) from home, but will not receive biofeedback training. Each session is expected to last 30 minutes to allow for completion of questionnaires over the the phone prior to and following each training session.

It is hypothesized that the biofeedback intervention will demonstrate high feasibility and compared to those in the control group, participants who receive the biofeedback intervention will attain greater pre-post reductions in both physiological and self-reported stress.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65
* Diagnosis of tetraplegia with residual sensory or motor impairments
* Discharged from inpatient rehabilitation and living in the community
* Access to high-speed internet at home
* Willingness to download the videoconferencing software Zoom
* Access to a mobile phone and willingness to download HRV software

Exclusion Criteria:

* Does not speak English
* Scores less than 37 on the STAI
* Unable to travel to Craig for an initial assessment
* History of participating in biofeedback training
* Requires mechanical ventilation
* Dependent on diaphragm pacer for respiration
* Currently in treatment for anxiety (e.g., pharmacologic or psychotherapeutic)
* Associated medical condition for which biofeedback is contraindicated (e.g., psychosis, pacemaker, or other implantable electric device)
* Currently hospitalized for medical/rehabilitation treatment
* Unable to commit to the four-week intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change in physiological stress | Session #1 (week 1) and Session #8 (week 4)
  Average LF (ms2)
Change in Depression Anxiety Stress Scale-21 (DASS-21) scores | Baseline (week 0) and Session #8 (week 4)
  The Depression Anxiety Stress Scale-21 (DASS-21) is a self report instrument designed to measure core symptoms of depression, anxiety, and stress. Each of the three DASS-21 scales contains seven items, divided into subscales with similar content. Scores for depression, anxiety, and stress are calculated by summing the scores for the relevant items. Items are rated on a scale from 0 (did not apply to me at all) to 3 (applied to me very much or most of time), with higher scores indicating more depression, anxiety, and stress.
Change in Subjective Units of Distress Scale (SUDS) scores | Baseline (week 0) and Session #8 (week 4)
  The Subjective Units of Distress Scale (SUDS) is a single-item self report instrument designed to measure the intensity of feelings and other internal experiences such as anxiety, anger, agitation, stress, or other painful feelings. A scale of 0 to 100 will be used to measure the subjective intensity of disturbance or distress experienced by the participant. A higher score indicates greater distress.

SECONDARY OUTCOMES:
Symptom list | After intervention session #1 (week 1), before and after intervention sessions #2-8 (weeks 1 through 4)
  A list of self-reported symptoms will be used to track any new symptoms requiring medical attention that emerge during the course of the study.
State Trait Anxiety Inventory (STAI) | After intervention sessions #1-8 (weeks 1 through 4)
  The State Trait Anxiety Inventory (STAI) is a 40 item self-report inventory consisting of 20 items to assess trait anxiety and 20 items to assess state anxiety. Items are rated on a scale from 1 (not at all) to 4 (very much). A total score is calculated by summing all six scores, multiplying the sum by 20, and then dividing by six. Total scores range from 20 - 80 with higher scores indicating greater self-reported anxiety. A normal score on the STAI is 34 - 36.

OTHER OUTCOMES:
Brief Pain Inventory (BPI) - 4 pain severity items | Baseline (week 0) and Session #8 (week 4)
  The Brief Pain Inventory (BPI) is one of the most widely used tools to assess pain. For this study, the four pain severity items will be used to assess worst, least, average, and current pain.
Brief Pain Inventory (BPI) - current pain severity item | Before and after intervention Sessions #1-7 (weeks 1 - 3)
  A single item from the Brief Pain Inventory (BPI) will be used to assess the severity of current pain.
Brief Pain Inventory (BPI) - pain relief item | After each intervention Session #1-8 (weeks 1 - 4)
  A single item from the Brief Pain Inventory (BPI) has been modified from, "In the last 24 hours, how much relief have pain treatments or medications provided? Please mark the box below the percentage that most shows how much relief you have received" to read, "During this session, how much pain relief did you experience? Please indicate the percentage that best describes how much relief you received."
Impact of study participation | Session #8 (week 4)
  Impact of Study Participation is a single open-ended item used to determine if study participation impacted anything other than stress, anxiety, or pain. Following the final session, participants will be asked, "Are there conditions other than stress, anxiety, or pain that were impacted by your participation in this study? If so, please list."

CONTACTS AND LOCATIONS:
Locations (1):
- Craig Hospital, Englewood, Colorado, United States

REFERENCES:
- [Derived] Monden KR, Nupp J, Ali A, MacIntyre B, Sevigny M, Hanks Philippus A. Exploring the feasibility of heart rate variability biofeedback for individuals with tetraplegia: A pilot clinical trial. Rehabil Psychol. 2025 May;70(2):214-225. doi: 10.1037/rep0000577. Epub 2024 Sep 9. PMID 39250283